CLINICAL TRIAL: NCT07267091
Title: The Burden of Lupus in Canada From a Patient Perspective: A Canadian Real-World PROxy Study
Status: Completed | Type: Observational
Sponsor: PeriPharm (Other)
Responsible Party: Sponsor
Other Study IDs: PROxy250918
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lupus; Lupus Arthritis; Lupus Arthritis, Systemic Lupus Erythematosus; Quality of Life (QOL)
Keywords: lupus; quality of life; real-world
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lupus: Adult patients with lupus member of Lupus Canada database
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No specific intervention is assess in this study. Observational cohort.

SUMMARY:
This study aims to capture the Canadian patient experience, burden, barriers, and treatment preferences. The findings will generate real-world evidence to support patient-centered care and guide healthcare providers, researchers, and decision-makers in improving support and treatment for people living with lupus.

DETAILED DESCRIPTION:
Lupus Canada will distribute an invitation to participate in the study through their mailing list, website, social networks providing a link to the questionnaire. Their mailing list database comprises about 8,000 individuals, including patients. Lupus Canada will reach out to the lupus community to inform them about their eligibility to participate in the study. Those meeting the eligibility criteria will be invited to sign the informed consent form (ICF) and complete all the study questionnaires on the PROxy web-based platform. For any questions, interested participants will have access to the contact information of the PROxy team, and a designated team member will communicate with participants by phone to answer all questions.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Part of the Lupus Canada database;

   a. Self-identified as a patient with Lupus.
3. Ability to read and understand English or French;
4. Signature of informed consent form.

Exclusion Criteria:

1. Participation in an interventional clinical trial for Lupus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Lupus who are part of Lupus Canada database
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
To estimate quality of life of patients with lupus | At recruitment
  Using the 36-item Short Form (SF-36) questionnaire, a generic health-related quality of life questionnaire containing 8 domains. Each domains score ranges from 0 to 100, where 0 represents poor health and 100 best possible health.

SECONDARY OUTCOMES:
To estimate work productivity impairment of patients with lupus. | At recruitment
  Using the Work Productivity and Activity Impairment (WPAI) questionnaire.
  This questionnaire provides a quantitative measure of impairment over the last 7 days and includes four metrics: absenteeism (work time missed because of health issues during the past 7 days), presenteeism (impairment while working due to health issues during the past 7 days), overall work productivity loss (combination of absenteeism and presenteeism), and activity impairment.
Indirect Costs and Patients' Preference Questionnaire | At recruitment
  Using a self-administered, 19-item questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- PROxy Network, an initiative of PeriPharm Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No